CLINICAL TRIAL: NCT02033837
Title: Evaluation of Cardiac CT Appropriateness at Second-generation 320-row CT With 0.275-sec Gantry Rotation Speed
Brief Title: Evaluation of Cardiac CT Appropriateness at Second-generation 320-row CT
Status: Completed | Type: Observational
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Daisuke Utsunomiya, Lecturer, Kumamoto University
Other Study IDs: Kuma1594
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Coronary Artery Disease; Cardiac CT
Keywords: Coronary artery disease; Cardiac CT; Appropriate Use Criteria (AUC)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
The influence of the second-generation 320-row area-detector CT (ADCT) on the clinical indications and appropriateness of cardiac CT has not been adequately investigated. The purpose of the survey is to assess the distribution of appropriateness ratings and test outcomes of cardiac CT with second-generation ADCT.

ELIGIBILITY:
Inclusion Criteria:

* indicated for coronary CT assessment

Exclusion Criteria:

* aortic disease
* pulmonary embolism
* severe arrhythmia
* severe heart failure
* allergy for iodinated contrast agent

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred for coronary CT angiography at our hospital
Sampling Method: Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2013-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
significant coronary stenosis | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Kumamoto University, Kumamoto, Japan